CLINICAL TRIAL: NCT03939546
Title: The FOUNDATION Study: Hospital Formulation Of B. Infantis EVC001 Utilized In The NICU To Demonstrate Tolerability In The Investigator's Preterm Neonates
Brief Title: The FOUNDATION Study
Acronym: FOUNDATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: EV-8801
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, prospective, cohort study. A prospective control cohort of 15 infants will initially be enrolled. Fifteen (15) infants will then be enrolled into the B. infantis cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Control Arm will not receive any study intervention or placebo. The infants in this arm will receive standard NICU care.
- B. infantis EVC001 (Active Comparator): Infants in the B. infantis arm will receive a once daily enteral feed of Evivo with MCT oil (8B CFU B. infantis EVC001) from Study Day 0 (by Day 10 of life) to hospital discharge, except on days when the infant is NPO.
  Interventions: Other: B. infantis EVC001

INTERVENTIONS:
Other: B. infantis EVC001 — Bifidobacterium longum subspecies infantis strain EVC001, designated a "Foods for Special Dietary Use" (FSDU)
  Other Names: Evivo with MCT Oil
  Arms: B. infantis EVC001

SUMMARY:
The FOUNDATION study will evaluate the tolerability of feeding preterm infants a B. infantis probiotic (EVC001) as the primary endpoint. This particular strain of Bifidobacterium has been shown to uniquely utilize oligosaccharides found in human breast milk, possibly providing a nutritional benefit for the infant consuming breast milk when B. infantis is colonized in the gut.

DETAILED DESCRIPTION:
This is a single-center, open-label, prospective, cohort study of an infant probiotic (Food for Special Dietary Use) conducted in the neonatal intensive care unit (NICU). Each subject enrolled will be in the study from the time of consent (within 10 days of birth) to hospital discharge. A prospective control cohort of 15 infants will initially be enrolled. Fifteen (15) infants will then be enrolled into the B. infantis cohort. Infants in the B. infantis cohort will receive a daily feeding of B. infantis EVC001 in MCT oil until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight < 1500 grams or gestational age at birth < 33 and 0/7 weeks
2. ≤ 10 days of life and considered viable
3. Consuming exclusive human milk diet (mother's milk or donor milk) with or without fortifier at time of enrollment
4. Toleration of 1.0 mL bolus enteral feeds

Exclusion Criteria:

1. Presence of septicemia or active infection as determined by positive 48-hour blood cultures
2. Necrotizing enterocolitis
3. Pulmonary hypoplasia
4. Presence of clinically significant congenital heart disease or other major congenital malformation
5. Any infant the Investigator deems to be ineligible for participation

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Tolerability: Frequency of Adverse Events | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by Adverse Events. Frequency of treatment-emergent adverse events (TEAEs), serious TEAEs and TEAEs causing premature discontinuation will be provided by treatment group.
Tolerability: Frequency of Probiotic Sepsis, as determined by the Principal Investigator | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by Probiotic Sepsis, as diagnosed by the PI. Frequency of Probiotic Sepsis will be provided by treatment group.
Tolerability: Frequency of Blood in Stool | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by visualized frank blood in stool. Frequency of blood in stool will be provided by treatment group.
Tolerability: Frequency of Abdominal Distension | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by abdominal distension causing treatment, diagnostics, or change in institutional standard of care. Frequency of abdominal distension will be provided by treatment group.
Tolerability: Frequency of Emesis | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by significant or bilious emesis causing treatment, diagnostics, or change in institutional standard of care. Frequency of emesis will be provided by treatment group.
Tolerability: Frequency of disruption in skin integrity in diaper area | From the time of study product administration through study completion, which occurs at the time of hospital discharge. Anticipated length of stay for this patient population is up to 84 days.
  Tolerability of B. infantis EVC001 in preterm infants as determined by disruption in skin integrity in diaper area requiring treatment. Frequency of disruption in skin integrity will be provided by treatment group.

SECONDARY OUTCOMES:
B. infantis levels in preterm infant stool related to probiotic supplementation | Baseline; Study Days 14 and 28; and 34, 36, and 38 weeks gestational age
  Effect of B. infantis EVC001 on the gut microbiome of preterm infants. DNA will be extracted from stool swab samples and will be used for quantitative PCR to determine levels of B. infantis.
Bifidobacterium levels in preterm infant stool related to probiotic supplementation | Baseline; Study Days 14 and 28; and 34, 36, and 38 weeks gestational age
  Effect of B. infantis EVC001 on the gut microbiome of preterm infants. DNA will be extracted from stool swab samples and will be used for quantitative PCR to determine levels of Bifidobacterium.
Changes in the preterm gut microbiome over time related to probiotic supplementation | Baseline; Study Days 14 and 28; and 34, 36, and 38 weeks gestational age
  Effect of B. infantis EVC001 on the gut microbiome of preterm infants. DNA and RNA will be extracted from stool swab samples and will be used for next generation sequencing to determine relative abundance of the most abundant bacterial taxa.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bajorek, MD, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health Winnie Palmer Hospital for Women & Babies, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No